CLINICAL TRIAL: NCT01276834
Title: Randomised Comparison of Two Different Immunosuppressive Regimens on Progression of Arteriosclerosis in Renal Transplant Patients.
Brief Title: Comparison of Immunosuppression on Progression of Arteriosclerosis in Renal Transplantation
Acronym: NOCTX-2
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient patients enrolled
Sponsor: Dianet Dialysis Centers (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Principal Investigator, B.C. van Jaarsveld, MD PhD, MD, PhD, Dianet Dialysis Centers
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOCTX-2; 2009-011605-16 (EudraCT Number)
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Renal Transplantation
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- everolimus-based immunosuppression (Experimental): immunosuppression with everolimus, prednisone and mycophenolate
  Interventions: Drug: everolimus
- standard immunosuppression (Active Comparator): immunosuppression with tacrolimus, prednisone and mycophenolate
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus — comparison of everolimus-based and CNI-based immunosuppression

SUMMARY:
To compare in a prospective randomised way the effect of two different immunosuppressive regimens - mTOR-based regimen or CNI-based regimen - on the progression of coronary artery calcification in renal transplant patients measured at baseline, 1, 2, and 3 years after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-75 yr
* Willingness to provide written informed consent
* Ability to understand the study procedures

Exclusion Criteria:

* Life expectancy < 3 months
* Claustrophobia
* Allergy to iodinated contrast
* Treatment incompliance
* Pregnancy
* Highly HLA-sensitized patients
* Severe dyslipidemia or proteinuria
* Severe leucopenia or thrombocytopenia
* GFR < 30 ml/min

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
change in coronary artery calcification score | 3 years
  Comparison in a randomised way the effect of a calcineurin-based immunosuppressive regimen with an mTOR-based regimen on progression of coronary calcification on renal transplant patients.
  The results of this study will provide more insight in protection against cardiovascular disease in renal transplant patients.

CONTACTS AND LOCATIONS:
Overall Officials: Franka E van Reekum, MD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands